CLINICAL TRIAL: NCT06068803
Title: Investigating the Immunometabolic and Cognitive Effects of 4 Weeks of Ketone Supplementation in Older Adults
Brief Title: Do Ketone Drinks Improve Immune, Metabolic and Cognitive Health in Older Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Anna Nicholas, Principal Investigator, University of Bath
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 23/SW/0067
Record Dates: First submitted 2023-09-13; First posted 2023-10-05 (Actual); Last update posted 2023-10-05 (Actual); Status verified 2023-09

CONDITIONS: Aging
Keywords: Ketone
MeSH Terms: conditions — Ketosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketone drink (Experimental): Pre-intervention (baseline) and post-intervention measurements will be obtained before and after the 4-week supplementation period. Physical activity and blood glucose will be monitored using wearable devices.
  Interventions: Dietary Supplement: Ketone drink
- Placebo (Placebo Comparator): Pre-intervention (baseline) and post-intervention measurements will be obtained before and after the 4-week supplementation period. Physical activity and blood glucose will be monitored using wearable devices.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Ketone drink — Participants will consume three daily ketone monoester (KME) drinks (0.282g KME/kg body weight/ serving) for 4 weeks.
  Other Names: D-β-hydroxybutyrate-R 1,3-Butanediol
  Arms: Ketone drink
Dietary Supplement: Placebo — Participants will consume three daily taste-matched calorie-free placebo drinks for 4 weeks.
  Arms: Placebo

SUMMARY:
The goal of this randomised, double-blinded, placebo-controlled trial is to investigate the immune, metabolic and cognitive effects of four weeks of daily ketone supplementation in adults aged 60 to 80 with stable health. The main objectives are to assess the effects of the intervention versus placebo on markers of metabolic health, inflammation, immune function, adipose tissue, and cognitive performance.

Participants will undergo two weeks of baseline monitoring followed by a four-week supplementation period in which they will drink a ketone monoester drink or taste-matched placebo three times a day. During these periods, participants will record their diet and supplement intake and their physical activity and blood glucose will be monitored using wearable devices. At the beginning and end of the supplementation period, participants will undergo testing in the university physiology laboratories, involving blood, expired air and adipose tissue samples, as well as cognitive tests, physical tests and questionnaires.

DETAILED DESCRIPTION:
Background: Research shows that ketones have beneficial effects on metabolism, inflammation and brain health in humans. In mice, they have also been shown to influence pathways involved in ageing. Ketones are natural molecules that are produced by the body when people fast (abstain from eating) for longer than 16-24 hours or eat a diet low in carbohydrates. It is now possible to consume ketones in the form of a drink.

Aims: This study aims to investigate if consuming a ketone drink for four weeks improves immunometabolic and cognitive health in adults aged 60 to 80 years. The main objectives are to assess the effects of the intervention versus placebo on:

1. Markers of metabolic health, including glucose control, lipid profile, blood pressure and body composition;
2. Systemic inflammation, immune cell activation and pro-inflammatory cytokine production;
3. Gene expression and secretory profile of subcutaneous adipose tissue; and
4. Cognitive performance and physical function.

Methods: The study is a randomised, double-blinded, placebo-controlled trial. Thirty participants (male and female) aged 60 to 80 years old with stable health will be recruited. Participants will undergo two weeks of baseline monitoring followed by a four-week supplementation period in which they will drink a ketone monoester drink or placebo three times a day. During these periods, participants will record their diet and supplement intake and their physical activity and blood glucose will be monitored using wearable devices. For two days in the supplementation period, participants will replicate their food consumption and physical activity so that they match two days in the baseline period (these are known as matched meal and activity days).

At the beginning and end of the supplementation period, participants will come to the physiology laboratories at the University of Bath for testing. Here, measures will be taken of their body weight, body composition, blood pressure, cognitive function and physical function, as well as samples of expired air, fat tissue and blood for analysis. Sleep and quality of life will be assessed via questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Age 60 to 80 years
* Postmenopausal women must be >1 year since last menses
* Able to provide informed consent
* Willing and able to comply with all study procedures including randomisation into any of the experimental groups; maintenance of habitual dietary intake, exercise, medication and supplement use over the 28-day intervention period; blood draws and adipose tissue biopsies; and abstinence from alcohol (>24 h), food (>10 h) and strenuous exercise (>3 d) prior to trial days.

Exclusion Criteria:

* Living in a residential care home
* Unstable or clinically active pulmonary, cardiac, hepatic, renal, endocrine, hematologic, immunologic, neurologic, psychiatric or biliary disorders. 'Unstable' refers to complications of a condition that are not controlled by medication or lifestyle and which require frequent monitoring and testing by a health professional. Stable chronic disease is not an exclusion criterion unless specified.
* Diagnosed Type 1 or Type 2 Diabetes Mellitus
* Diagnosed gastrointestinal condition which would potentially impact ability to consume study drink (e.g. inflammatory bowel disease, history of gastrointestinal ulcers or bleeding)
* Diagnosed autoimmune condition
* Previous major cardiovascular event (e.g. heart attack, stroke)
* Past or current cancer diagnosis and treatment excluding non-melanoma skin cancers
* Severe hypertension (systolic blood pressure ≥180 mmHg and/or diastolic blood pressure ≥120 mmHg), as defined by blood pressure measured at Visit 1
* Current tobacco or recreational drug use
* Reported changes to use of thyroid, antihypertensive, antidepressant or statin medications within 30 days of Visit 1
* Taking medications that will interfere with the study outcomes
* Known negative reaction to lidocaine anaesthetic and/or taking warfarin
* Currently following a ketogenic diet or taking ketone supplements
* Not weight stable in the prior 3 months (>5% weight change)
* Unable to converse in English

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-14 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in 24hr average glucose area under the curve (AUC) | 1 day during baseline period and 1 day during the intervention period
  Glucose control will be measured using a continuous glucose monitoring device worn throughout the baseline period and weeks 3 and 4 of the intervention period. Change in 24h average glucose AUC will be assessed on 'matched meal and activity days' i.e. days during intervention and baseline that are matched for food intake and physical activity.

SECONDARY OUTCOMES:
Change in glycemic variability | 1 day during baseline period and 1 day during the intervention period
  Glucose control will be measured using continuous glucose monitoring device worn throughout the baseline period and weeks 3 and 4 of the intervention period. Change in glycemic variability will be assessed on 'matched meal and activity days' i.e. days during intervention and baseline that are matched for food intake and physical activity.
Change in serum fructosamine | Pre (day 0) and post (day 29)
  Measured in fasting blood sample by automated analyser (Daytona Rx)
Change in fasting plasma glucose | Pre (day 0) and post (day 29)
  Measured in fasting blood sample by automated analyser (Daytona Rx)
Change in fasting lipid profile concentrations | Pre (day 0) and post (day 29)
  Measured in fasting blood sample by automated analyser (Daytona Rx)
Change in fasting plasma free fatty acids (FFA) | Pre (day 0) and post (day 29)
  Measured in fasting blood sample by automated analyser (Daytona Rx)
Change in fasting plasma insulin | Pre (day 0) and post (day 29)
  Measured in fasting blood sample using a high-sensitivity human insulin enzyme-like immunosorbent assay (ELISA)
Change in Insulin Sensitivity Index | Pre (day 0) and post (day 29)
  Calculated from fasting plasma insulin and fasting plasma glucose
Change in Adipose tissue Insulin Resistance index (Adipo-IR) | Pre (day 0) and post (day 29)
  Calculated from fasting plasma insulin and fasting plasma FFA
Change in body mass | Pre (day 0) and post (day 29)
  Measured using a digital body weight scales
Change in waist and hip circumference | Pre (day 0) and post (day 29)
  Measured using a measurement tape
Change in waist to hip ratio | Pre (day 0) and post (day 29)
  Calculated from waist and hip circumferences
Change in fat mass and fat free mass | Pre (day 0) and post (day 29)
  Assessed by Dual Energy X-ray Absorptiometry (DEXA) scan
Change in calf muscle density, quality and area | Pre (day 0) and post (day 29)
  Assessed by calf peripheral Quantitative Computed Tomography (pQCT)
Change in blood pressure | Pre (day 0) and post (day 29)
  Measured using an automated blood pressure device. Both systolic and diastolic blood pressure will be measured
Change in circulating adipokines and inflammatory cytokines | Pre (day 0) and post (day 29)
  Key inflammatory cytokines including CRP will be quantified by R-plex, U-plex and V-plex kits on a Mesoscale QuickPlex SQ120
Change in blood immune cell phenotype, function and activation | Pre (day 0) and post (day 29)
  Peripheral blood mononuclear cells (PBMCs) isolated from whole blood will be incubated with fluorophore-conjugated antibodies and analysed with a flow cytometer to examine the phenotype and cytokine production of immune cells
Change in adipose tissue immune cell phenotype, function and activation | Pre (day 0) and post (day 29)
  Adipose tissue stromal vascular fraction (SVF) will be incubated with fluorophore-conjugated antibodies and analysed with a flow cytometer to examine the phenotype and cytokine production of immune cells
Change adipose tissue adipokine and cytokine concentrations | Pre (day 0) and post (day 29)
  Adipose tissue explants will be cultured ex vivo for 3h. Concentrations of key adipokines and cytokines in supernatant will be quantified by R-plex, U-plex and V-plex kits on a Mesoscale QuickPlex SQ120
Change in adipose tissue gene expression | Pre (day 0) and post (day 29)
  Whole-tissue RNAseq
Change in Digit-Symbol Substitution Test score | Pre (day 0) and post (day 29)
  This test will be administered using the computer-based app Inquisit6 Lab (Millisecond). The score reflects the number of correct symbols within the allowed time. Higher is better.
Change in Stroop Test score | Pre (day 0) and post (day 29)
  This test will be administered using the computer-based app Inquisit6 Lab (Millisecond). The score reflects the number of correct responses and the response latency. Higher is better.
Change in Trail Making Task score | Pre (day 0) and post (day 29)
  This test will be administered using the computer-based app Inquisit6 Lab (Millisecond). The score reflects the time taken to complete trails A and B. Lower is better.
Change in Digit Span Test score | Pre (day 0) and post (day 29)
  This test will be administered using the computer-based app Inquisit6 Lab (Millisecond). The score reflects the maximum number of digits recalled correctly. Higher is better.
Change in score on Montreal Cognitive Assessment (MoCA) | Pre (day 0) and post (day 29)
  The test will be administered by a trained researcher.

OTHER OUTCOMES:
Change in physical activity level (PAL) | Pre (day 0) and post (day 29)
  Physical activity will be assessed using a combined accelerometer and heart rate monitor (Actiheart) worn throughout the baseline period and weeks 3 and 4 of the intervention period
Change in heart rate | Pre (day 0) and post (day 29)
  Heart rate will be assessed using an accelerometer (Actiheart) worn throughout the baseline period and weeks 3 and 4 of the intervention period
Change in score on Pittsburgh Sleep Quality Index | Pre (day 0) and post (day 29)
  Questionnaire to assess sleep quality
Change in score on EuroQuol EQ-5D-5L Questionnaire | Pre (day 0) and post (day 29)
  Questionnaire to assess health-related quality of life
Change in Short Physical Performance Battery score | Pre (day 0) and post (day 29)
  Standard set of tests to measure physical function in elderly involving gait speed, chair stand and balance test
Supplement acceptability as assessed by likability, taste and ease of compliance | Post (day 29)
  Acceptability of the supplement will be assessed via questionnaire using a 7-point Likert scale
Change in adipose tissue protein expression | Pre (day 0) and post (day 29)
  Adipose tissue protein expression will be assessed by targeted immunoblotting.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: No